CLINICAL TRIAL: NCT04863274
Title: The Program to Assess the Influence of Routing and In-depth Consultation of Patients With Cardiovascular Risk Factors on the Choice of Medicine and Treatment Compliance
Brief Title: Influence of Additional Physician's Consultations and Short Message Service (SMS) Reminders to Patient Compliance
Acronym: 3P
Status: Completed | Type: Observational
Sponsor: The League of Clinical Research, Russia (Other)
Collaborators: National Research Center for Preventive Medicine (Other Government)
Responsible Party: Sponsor
Other Study IDs: Primary Prevention Program
Record Dates: First submitted 2021-01-20; First posted 2021-04-28 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-04

CONDITIONS: Lipid Metabolism Disorders
Keywords: prevention of cardiovascular diseases; atorvastatin
MeSH Terms: conditions — Lipid Metabolism Disorders | interventions — Atorvastatin; Spermine Synthase

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Expanded consultation group: In an expanded consultation group is being conducted in the study group on the importance of primary prevention of cardiovascular diseases and on the reduction of cardiovascular risk by taking statins. Patients are given brochures and information materials on the risk factors for cardiovascular diseases and the possibility of their correction. Also, the patients of the study group are regularly reminded (2 times a month) with the help of SMS mailings and calls of health workers about the need to follow the doctor's recommendations for taking atorvastatin and returning to the medical institution.
  Interventions: Drug: atorvastatin

INTERVENTIONS:
Drug: atorvastatin — Profound patients' consultations (different from standard practice) on the importance of primary prevention of cardiovascular diseases, including preventive administration of statins.
  Subjects in profound consultation group will receive regular reminders (2 times a month) via SMS and phone calls to check following the doctor's recommendations and remind about follow-up visit to study centre.
  Other Names: SMS and phone call reminders; Patients' consultations

SUMMARY:
A systematic collection of retrospective and prospective data based on non-interventional patient observation, aimed to assess the risks, course and outcomes of a disease or a group of diseases:

* the retrospective part: database of patients with cardiovascular risks;
* the prospective part: observation of patients in the real world medical practice.

DETAILED DESCRIPTION:
The research program will have two parts:

Stage 1: identification of patients with moderate, high and very high cardiovascular risk, not having diseases of atherosclerotic genesis and requiring lipid-lowering drugs.

Stage 2: a prospective observation of patients receiving primary medical prophylaxis of CVD with atorvastatin.

ELIGIBILITY:
Inclusion criteria:

Data on the following subjects is planned to be collected in the project:

* Aged from 40 to 65 years inclusively
* With a high (≥5%) cardiovascular risk measured by SCORE and low density lipoprotein (LDL) levels of ≥2,5 mmol/L, or with a very high (≥10%) cardiovascular risk measured by SCORE and LDL levels ≥1,8 mmol/L or With atherosclerotic stenosis of brachiocephalic arteries of >50% in the absence of cerebrovascular disease

Exclusion criteria:

* No contraindications to statin treatment and not taking stating at study entry.
* History of the following clinically significant events and conditions:

  (а) myocardial infarction (б) stroke (в) transient ischemic attack
* Presence of the following diseases at the time of a statin administration:

  (а) ischemic heart disease (б) heart failure (в) peripheral artery atherosclerosis (г) atherosclerotic stenosis of brachiocephalic arteries with cerebrovascular disease .

Subjects must give their consent for processing of their personal data for the purposes of this scientific project.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The total population of patients (2912 people) will be divided into three strata:
  patients with moderate risk of CVD (1242 patients) patients with high risk of CVD (1044 patients) patients with very high risk of CVD (626 patients). The subjects are randomized to a study or control group in each stratum in the ratio of 1: 1
Sampling Method: Probability Sample
Enrollment: 2912 (Actual)
Dates: Start 2018-06-21 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
Target level of LDL cholesterol | 12 months
  To assess number of patients achieving the target level of low-density lipoprotein cholesterol in study group and in control group.

CONTACTS AND LOCATIONS:
Overall Officials: Svetlana I Elkonina, MD, Study Director — League of Clinical Research (LeagueCRR)
Locations (1):
- League of Clinical Research (LeagueCRR), Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2018-03-30): https://cdn.clinicaltrials.gov/large-docs/74/NCT04863274/Prot_000.pdf